Ethiodized oil-based chemoembolization for hepatocellular carcinoma: Randomized

controlled trial of aqueous cisplatin emulsion versus anhydrous cisplatin suspension

Date: 16 July 2016

Statistical analysis

Efficacy analyses are performed on the per-protocol population according to the treatment

finally received with adherence to the protocol. Post-randomization exclusion is limited only

to those who withdrew themselves from the study or who have not completed the required

treatments. For continuous variables, median with inter-quarter range (IQR) are provided and

compared using U test between the groups. For dichotomic variables, comparison between

groups is performed using Chi-square test or Fisher's exact test. The time-to-event data in

months are estimated with the method of Kaplan-Meier analysis for TTP, PFS and OS, and

presented with median and 95% confidence interval (CI). If the median is not reached, 3-year

and 5-year rate are given. Survival outcomes between the groups are compared using log-rank

test, hazard ratio (HR) and corresponding 95% confidence interval (CI) are computed using

cox regression model. SPSS software is used for analysis. Statistical significance is p< 0.05.